CLINICAL TRIAL: NCT03692091
Title: Comparing Two Methods of Subacromial Space Injection - A Randomised Blinded Trial
Brief Title: Comparing Two Methods of Subacromial Space Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aneurin Bevan University Health Board (Other)
Responsible Party: Principal Investigator, Vasantha Kumar Ramsingh, Locum Consultant Orthopaedic Surgeon, Aneurin Bevan University Health Board
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRAS194489
Record Dates: First submitted 2018-09-03; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior portal (Active Comparator): Injection in to subacromial space from anterior portal
  Interventions: Procedure: Subacromial Injection
- Lateral portal (Active Comparator): Injection in to subacromial space from lateral portal
  Interventions: Procedure: Subacromial Injection

INTERVENTIONS:
Procedure: Subacromial Injection — Injection in to subacromial space in the shoulder from anterior portal

SUMMARY:
Subacromial shoulder injections can be approached from the front or side of the shoulder. The investigators are comparing both methods, to find which one has better spread in the subacromial space.

DETAILED DESCRIPTION:
Both lateral and posterio-lateral methods of subacromial injections are widely used for diagnostic and therapeutic purposes. It is not known which method allows the most accurate access into the subacromial space and is more effective.

The investigators have been using a novel approach from the anterior aspect of the shoulder for years with good clinical effect and propose comparing this approach to the described approach. This study will indicate which method is best and will be of practical clinical importance. The investigators feel the technique is easier to perform than other described methods and could be taught to clinicians throughout the country and adopted as the standard approach.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain for at least 6 weeks duration along the lateral aspect of the shoulder.
* Positive impingement signs.

Exclusion Criteria:

* History of compensation claim due to shoulder problems.
* Allergy to radiographic dye.
* Recent shoulder fracture.
* Bleeding disorder.
* Previous shoulder surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
The spread of dye in subacromial space | With in One hour
  The participants will go for an X ray following injection which contains a radio-opaque dye to demonstrate the spread of injected material (Local anaesthetic, depomedrone and Niopam dye) in the subacromial space. A blinded radiologist will read the radiographs and scale the distribution of dye from 1 to 4 depending on the location of radiopaque dye.

SECONDARY OUTCOMES:
Pain control after subacromial injection | With in One hour
  The participants will fill a visual analog score before and after injection to assess the pain relief after injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Aneurin Bevan University Health Board, Newport, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eustace JA, Brophy DP, Gibney RP, Bresnihan B, FitzGerald O. Comparison of the accuracy of steroid placement with clinical outcome in patients with shoulder symptoms. Ann Rheum Dis. 1997 Jan;56(1):59-63. doi: 10.1136/ard.56.1.59. PMID 9059143
- [Background] Calis M, Akgun K, Birtane M, Karacan I, Calis H, Tuzun F. Diagnostic values of clinical diagnostic tests in subacromial impingement syndrome. Ann Rheum Dis. 2000 Jan;59(1):44-7. doi: 10.1136/ard.59.1.44. PMID 10627426
- [Result] Yamakado K. The targeting accuracy of subacromial injection to the shoulder: an arthrographic evaluation. Arthroscopy. 2002 Oct;18(8):887-91. doi: 10.1053/jars.2002.35263. PMID 12368787
- [Result] Partington PF, Broome GH. Diagnostic injection around the shoulder: hit and miss? A cadaveric study of injection accuracy. J Shoulder Elbow Surg. 1998 Mar-Apr;7(2):147-50. doi: 10.1016/s1058-2746(98)90226-9. PMID 9593094